CLINICAL TRIAL: NCT00838305
Title: Role of Serotonin in Acute and Subacute MDMA Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 28.065-1
Record Dates: First submitted 2009-01-23; First posted 2009-02-06 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: MDMA Mechanism of Action
Keywords: MDMA; citalopram; serotonin; psychedelic
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): drug: placebo subjects also get citalopram and placebo in a 2x2 crossover design
  Interventions: Drug: Placebo
- mdma (Experimental): drug: mdma subjects also get citalopram and placebo in a 2x2 crossover design
  Interventions: Drug: MDMA and citalopram

INTERVENTIONS:
Drug: MDMA and citalopram — MDMA 1.5 mg/kg and citalopram 20 mg
  Arms: mdma
Drug: Placebo — drug: placebo subjects also get citalopram and placebo in a 2x2 crossover design
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the effects of MDMA (particularly its emotional effects) and to determine the role of serotonin in these effects. Serotonin is a neurotransmitter, which is a chemical that is released by some brain cells to communicate with other brain cells. Many of the effects of MDMA are thought to be the result of increased serotonin release.

In order to understand the effects of MDMA and role of serotonin in these effects, we will administer MDMA alone and in combination with the antidepressant citalopram (one trade name for this is Celexa). Citalopram decreases the ability of MDMA to release serotonin. Citalopram will therefore decrease any of MDMA's effects that are the result of serotonin release; we want to measure this.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 50 years
* Experienced with MDMA

Exclusion Criteria:

* Significant physical or psychiatric illness which might impair the ability to safely complete the study or that might be complicated by the study drugs, including prior seizures (after age 8), history of major depression, or other active neurological disease or clinically significant abnormalities on physical examination or screening laboratory values

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine if administration of the selective serotonin reuptake inhibitor (SSRI) citalopram decreases the subacute (post 24hr) discontinuation effects of MDMA in experienced MDMA users given a modest dose of MDMA | 24 hours

SECONDARY OUTCOMES:
To determine if administration of the SSRI citalopram decreases the acute (post 1 to 4hr) social and emotional and cognitive effects of MDMA | post 1-4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CPMC Research Institute, St.Luke's Hospital, San Francisco, California, United States